CLINICAL TRIAL: NCT00719394
Title: Ascending Single-Dose Study of the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of GSI-136 Administered Orally to Healthy Japanese Male Subjects and Healthy Japanese Elderly Male Subjects
Brief Title: Study Evaluating Safety of GSI 136 in Young and Elderly Japanese Males
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Wyeth (Registry Contact: Clinical Trial Registry Specialist), Wyeth
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 3225A1-1001
Record Dates: First submitted 2008-07-17; First posted 2008-07-21 (Estimated); Last update posted 2009-07-10 (Estimated); Status verified 2009-07

CONDITIONS: Alzheimer Disease; Healthy
Keywords: alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- GSI 136 (Experimental)
  Interventions: Drug: GSI 136
- placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: GSI 136
  Arms: GSI 136
Drug: placebo
  Arms: placebo

SUMMARY:
This is a first-in-human study of GSI-136, a gamma-secretase inhibitor being developed for the treatment of Alzheimer disease. This study will take place in Japan only and will provide an initial assessment of the safety, tolerability, pharmacokinetics (PK), and pharmacodynamics (PD) of GSI-136 after administration of ascending single oral doses to healthy Japanese male subjects and healthy Japanese elderly male subjects.

ELIGIBILITY:
Inclusion Criteria .

1. Men aged 20 to 45 years, or greater than 65 years, inclusive, at screening and who agree to use a medically acceptable form of contraception during the study and to continue its use for 12 weeks after test article administration.
2. Healthy as determined by the investigator on the basis of medical history, physical examination, clinical laboratory tests, vital sign measurements and 12-lead electrocardiogram (ECG).

Exclusion Criteria

1. Presence or history of any disorder that may prevent the successful completion of the study.
2. Any history or presence of chronic respiratory disorder or disease including but not limited to asthma, sleep apnea, or chronic obstructive pulmonary disease (COPD).

Min Age: 20 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2008-03; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of GSI-136 as evaluated from reported adverse events, scheduled physical examinations, vital sign measurements, orthostatic vital sign measurements, cardiac rhythm monitoring, 12-lead ECGs, and clinical laboratory test results. | 6 months

SECONDARY OUTCOMES:
Pharmacokinetics as evaluated from the blood and urine concentrations of GSI-136; Pharmacodynamics as evaluated from the levels of select biomarkers in the blood and the administration of a visual analog scale to measure sedation effects. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (1):
- Tokyo Heat Center, Tokyo, Japan